CLINICAL TRIAL: NCT03857542
Title: A Phase 3, Multicenter, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety and Efficacy of AGN-190584 in Participants With Presbyopia
Brief Title: A Phase 3 Efficacy Study of Pilocarpine HCl Ophthalmic Solution (AGN-190584) in Participants With Presbyopia
Acronym: GEMINI 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1883-302-013
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Results first posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vehicle (Placebo Comparator): Participants received one drop of vehicle in each eye, once daily, for up to 30 days.
  Interventions: Other: Vehicle
- Pilocarpine HCl Ophthalmic Solution (Experimental): Participants received one drop of pilocarpine HCl ophthalmic solution 1.25% in each eye, once daily, for up to 30 days.
  Interventions: Drug: Pilocarpine HCl Ophthalmic Solution

INTERVENTIONS:
Drug: Pilocarpine HCl Ophthalmic Solution — Pilocarpine HCl ophthalmic solution 1.25%, one drop in each eye, once daily, for up to 30 days.
  Other Names: AGN-190584; VUITY
  Arms: Pilocarpine HCl Ophthalmic Solution
Other: Vehicle — Vehicle, one drop in each eye, once daily, for up to 30 days.
  Arms: Vehicle

SUMMARY:
This clinical study will evaluate pilocarpine hydrogen chloride (HCl) ophthalmic solution (AGN-190584) in an expanded participant population to establish efficacy, safety, and tolerability versus the vehicle-control when administered, over a 30-day study intervention period, once daily bilaterally in participants with presbyopia.

ELIGIBILITY:
Inclusion Criteria

Subjective complaints of poor near vision that impact activities of daily living

Exclusion Criteria

Uncontrolled systemic disease

Any clinical condition or previous surgery that might affect the absorption, distribution, biotransformation, or excretion of AGN-190584. History of cataract surgery, phakic intraocular lens surgery, corneal inlay surgery, radial keratotomy, or any intraocular surgery. However, participants with history of photorefractive keratectomy (PRK) or laser-assisted in situ keratomileusis (LASIK) with corrected distance visual acuity (CDVA) meeting inclusion criteria will be allowed to enroll.

Known allergy or sensitivity to the study intervention or its components or other cholinergic agonist medications

Concurrent use of any topical ophthalmic medications, including artificial tears, other than the study intervention during the course of the study

Concurrent use of temporary or permanent punctal plugs or history of punctal cautery in one or both eyes

Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study

Participation in a blood or plasma donation program within 30 days prior to study intervention administration

Severe dry eye disease (defined as total corneal staining ≥ grade 3 on the 5-point Oxford scale and an ocular surface disease index (OSDI) score of > 33) at the screening visit

Corneal abnormalities (including keratoconus, corneal scar, Fuchs' endothelial dystrophy, guttata, or edema) in either eye that are likely to interfere with visual acuity

Narrow iridocorneal angles (Shaffer grade ≤ 2 or lower on gonioscopy examination), history of angle-closure glaucoma, or previous iridotomy

History of iris trauma, Adie's tonic pupil, abnormal pupil shape in either eye, or anisocoria > 1 mm between pupils under mesopic conditions at the screening visit

Lens opacity in either eye that is determined to cause significant disturbance of the central visual axis on screening biomicroscopy

Diagnosis of any type of glaucoma or ocular hypertension

Bifocal or multifocal spectacles or contact lenses for habitual correction. Participants willing to wear study-provided monofocal correction (either spectacles or contact lenses) during the study can be enrolled

Abnormal and clinically significant results according to the investigator or designee, on physical/ophthalmic examination or medical history

Females who are pregnant, nursing, or planning a pregnancy during the study

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 427 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Safyan, Study Director — Allergan
Locations (35):
- United States (35):
  - Eye Center South, Dothan, Alabama
  - M&M Eye Institute, Prescott, Arizona
  - Walman Eye Center, Sun City, Arizona
  - Milton M. Hom, OD, FAAO, Azusa, California
  - Global Research Management, Glendale, California
  - Advanced Vision Care, Los Angeles, California
  - North Valley Eye Medical Group, Inc., Mission Hills, California
  - Eye Research Foundation, Newport Beach, California
  - Corneal Consultants of Colorado, Littleton, Colorado
  - Benjamin Knox Lambright, MD, Crystal River, Florida
  - South Florida Vision Center, Fort Lauderdale, Florida
  - Bowden Eye Associates, Jacksonville, Florida
  - Mid Florida Eye Center, Mt. Dora, Florida
  - Newsom Eye & Laser Center, Sebring, Florida
  - Clayton Eye Center, Morrow, Georgia
  - The Midwest Center for Sight, Des Plaines, Illinois
  - Jacksoneye, Lake Villa, Illinois
  - Kannarr Eye Care, Pittsburg, Kansas
  - Heart of America Eyecare, Shawnee Mission, Kansas
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Chu Laser Eye Institute, Bloomington, Minnesota
  - Silverstein Eye Centers, Kansas City, Missouri
  - Moyes Eye Center, Kansas City, Missouri
  - Tekwani Vision Center, St Louis, Missouri
  - Amel Youssef, OD, Las Vegas, Nevada
  - Debry Medical Services PC, Las Vegas, Nevada
  - Bucci Laser Vision, Wilkes-Barre, Pennsylvania
  - Waring Vision Institute, Mt. Pleasant, South Carolina
  - University Eye Surgeons, Maryville, Tennessee
  - Total Eye Care, PA, Memphis, Tennessee
  - Keystone Research ltd. at Texan Eye, Austin, Texas
  - The Cataract and Glaucoma Center, El Paso, Texas
  - Texas Eye & Laser Ctr, Hurst, Texas
  - Benjamin Travis Dastrup, MD, Ogden, Utah
  - Vision Consultants and Surgeons, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Allergan will share de-identified patient-level data and study-level data including protocols and clinical study reports for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. More information can be found on http://www.allerganclinicaltrials.com/.
Supporting Information: Study Protocol, CSR
Time Frame: After having received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published.
Access Criteria: To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes.
URL: http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Distance-corrected near visual acuity (DCNVA) measurements at 1 site were not conducted correctly at the screening and baseline visits; all participants from this site were excluded from efficacy analyses.
Groups:
- Pilocarpine HCl Ophthalmic Solution: Participants received one drop of pilocarpine hydrochloride (HCl) ophthalmic solution 1.25% in each eye, once daily, for up to 30 days.
Period: Overall Study
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Started | 215 | 212
Completed | 209 | 207
Not Completed | 6 | 5
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Reason not Specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution | Total
Number analyzed (Participants) | 215 | 212 | 427
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (3.48) | 49.6 (3.71) | 49.8 (3.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 138 | 300
  Male | 53 | 74 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 37 | 78
  Not Hispanic or Latino | 174 | 175 | 349
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 35 | 64
  White | 176 | 171 | 347
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Gaining 3 Lines or More in Mesopic, High-contrast, Binocular DCNVA, Without Losing More Than 5 Letters of Mesopic, High-Contrast, Binocular CDVA With the Same Refractive Correction at Day 30, Hour 3
Description: Visual acuity for near (40 centimeter (cm)) and distance (4 meter (m)) targets were measured in mesopic conditions using an eye chart. High contrast corrected distance visual acuity (CDVA) was assessed binocularly (in each eye) using the provided visual acuity charts for distance vision in a room with mesopic lighting conditions measured at the target. Forced choice letter by-letter scoring was used for each test and the total number of correct letters or the highest value (number) of the grid identified (as applicable) were recorded. Mesopic condition was defined as low lighting 3.2 to 3.5 candelas per square meter (cd/m^2) measured at the target. DCNVA= distance-corrected near visual acuity.
Time Frame: Baseline (Day 1) to Day 30 (Hour 3)
Population: ITT Population included all randomized participants. Missing data was imputed as non-responders; excluding data from 1 site.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 203 | 196
percentage of participants | 10.8 | 26.0
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p < .0001, Chi-squared — P-value was adjusted for multiplicity control; Percentage Difference = 15.2, 95% CI 2-sided [7.7 to 22.7] — Analysis was done using Chi-square test. The 95% confidence intervals for the proportion differences were calculated based on the normal approximation based on pooled variance without continuity correction

2. Secondary Outcome: Percentage of Participants Gaining 3 Lines or More in Mesopic, High-contrast, Binocular DCNVA at Day 30, Hour 6
Description: Visual acuity for near (40 cm) target was measured in mesopic conditions using an eye chart. Mesopic condition was defined as low lighting 3.2 to 3.5 cd/m^2 measured at the target. Percentage of participants with 3 lines or more improvement from Baseline in mesopic, high-contrast DCNVA are reported.
Time Frame: Baseline (Day 1) to Day 30 (Hour 6)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 203 | 196
percentage of participants | 9.9 | 16.3
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0548, Chi-squared — P-value was adjusted for multiplicity control; Percentage Difference = 6.5, 95% CI 2-sided [-0.1 to 13.1] — Analysis was done using Chi-square test. The 95% confidence intervals for the proportion difference was calculated based on the normal approximation based on pooled variance without continuity correction

3. Secondary Outcome: Percentage of Participants Gaining 3 Lines or More in Mesopic, High-contrast, Binocular, DCNVA at Day 30, Hour 8
Description: Visual acuity for near (40 cm) was measured in mesopic conditions using an eye chart. Mesopic condition was defined as low lighting 3.2 to 3.5 cd/m^2 measured at the target. Baseline for efficacy was defined as the last non-missing efficacy assessment before the first dose of study intervention. Percentage of participants with 3 lines or more improvement from Baseline in mesopic, high-contrast DCNVA are reported.
Time Frame: Baseline (Day 1) to Day 30 (Hour 8)
Population: ITT Population included all randomized participants. Overall number of participants analyzed is the number of participants with data available for analysis at Baseline and timepoint; excluding data from 1 site.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 197 | 193
percentage of participants | 8.6 | 14.5
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0693, Chi-squared — P-value was adjusted for multiplicity control; Percentage Difference = 5.9, 95% CI 2-sided [-0.5 to 12.2] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in Mesopic, High-contrast, Binocular DCNVA Letters at Day 30, Hour 0.5
Description: Visual acuity for near (40 cm) target was measured in mesopic conditions using an eye chart. Mesopic condition was defined as lighting 3.2 to 3.5 cd/m^2 measured at the target. Mixed effect model for repeated measures (MMRM) was used for the analysis.
Time Frame: Baseline (Day 1) to Day 30 (Hour 0.5)
Population: ITT Population included all randomized participants. Overall number of participants analyzed is the number of participants with data available for analysis; excluding data from 1 site.
Measure: Least Squares Mean (Standard Error); unit: letters read correctly
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 197 | 193
letters read correctly | 4.7 (0.44) | 8.8 (0.44)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p < .0001, MMRM — MMRM with study intervention group, visit, visit by study intervention group interaction, age group, Baseline binocular DCNVA severity, iris color, emmetrope/non-emmetrope, Baseline value; Baseline value by visit interaction as fixed effects; P-value was adjusted for multiplicity control; Least Squares (LS) Mean Difference = 4.1, 95% CI 2-sided [2.9 to 5.2], Standard Error of Mean 0.59

5. Secondary Outcome: Percentage of Participants Achieving 20/40 or Better in Photopic, High-contrast, Binocular DCNVA at Day 30, Hour 1
Description: Visual acuity for near (40 cm) target was measured in photopic conditions using an eye chart. Photopic condition was defined as high lighting ≥80 cd/m^2 measured at the target.
Time Frame: Day 30 (Hour 1)
Population: ITT Population included all randomized participants. Overall number of participants analyzed is the number of participants with data available for analysis; excluding data for 1 site.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 198 | 193
percentage of participants | 82.8 | 92.7
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0141, Chi-squared — P-value was adjusted for multiplicity control; Percentage Difference = 9.9, 95% CI 2-sided [3.5 to 16.3] — Analysis was done using chi-square test. The 95% confidence intervals was calculated based on normal approximation based on pooled variance without continuity correction

6. Secondary Outcome: Mean Change From Baseline in Mesopic Near Vision Presbyopia Task-based Questionnaire (NVPTQ) Performance Score at Day 30, Hour 3
Description: NVPTQ had 12 questions on 4 reading tasks(reading a paragraph from book, excerpts from a newspaper article, portion of a nutrition label, and a section from restaurant menu). Participants completed specific reading tasks under mesopic conditions without any near-vision correction and answered 3 questions for each task, rated as 0=I could not read any text due to problems seeing up close,1=poor,2=fair,3=good,4=very good,5=excellent; impact of squinting as 0=No,I did not squint, 1=Yes, squinting helped me read some/all text, 2=Yes,but I still could not read any of the text; and satisfaction as 0=very dissatisfied to 4=very satisfied. The score based on vision-related ability and impact of squinting=(Book testlet+Newspaper testlet+Menu testlet+Nutrition Label testlet)/(testlets with non-missing responses), total possible score of 0-5. Higher scores=better outcomes;positive change from Baseline=improved performance (reading ability).
Time Frame: Baseline (Day 1) to Day 30 (Hour 3)
Population: ITT Population included all randomized participants. Overall number of participants analyzed is the number of participants with data available for analysis; excluding data for 1 site. ANCOVA was used for the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 197 | 192
score on a scale | 0.5 (0.09) | 1.3 (0.09)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p < .0001, ANCOVA — Analysis of covariance (ANCOVA) with study intervention group, age group, Baseline binocular DCNVA severity, iris color (brown/non-brown), emmetrope/non-emmetrope, and Baseline domain score as fixed effects; P-value was adjusted for multiplicity control; LS Mean Difference = 0.8, 95% CI 2-sided [0.5 to 1.0], Standard Error of Mean 0.12

7. Secondary Outcome: Change From Baseline in Photopic, High-contrast, Binocular Distance-corrected Intermediate Visual Acuity (DCIVA) Letters at Day 30, Hour 3
Description: Visual acuity for intermediate (66 cm) target was measured in photopic conditions using an eye chart. Photopic condition was defined as high lighting ≥80 cd/m^2 measured at the target. MMRM was used for the analysis.
Time Frame: Baseline (Day 1) to Day 30 (Hour 3)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: number of letters read correctly
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 198 | 193
number of letters read correctly | 2.9 (0.38) | 6.4 (0.39)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p < .0001, MMRM — MMRM with study intervention group, visit, visit by study intervention group interaction, age group, Baseline binocular DCNVA severity, iris color, emmetrope/non-emmetrope, Baseline value, and Baseline value by visit interaction as fixed effects; P-value was adjusted for multiplicity control; LS Mean Difference = 3.4, 95% CI 2-sided [2.4 to 4.4], Standard Error of Mean 0.52

8. Secondary Outcome: Percentage of Participants Gaining 3 Lines or More in Mesopic, High-contrast, Binocular, DCNVA at Day 30, Hour 10
Description: Visual acuity for near (40 cm) target was measured in mesopic conditions using an eye chart. Mesopic condition was defined as low lighting 3.2 to 3.5 cd/m^2measured at the target. Percentage of participants with 3 lines or more improvement from Baseline in mesopic, high-contrast, binocular DCNVA are reported.
Time Frame: Baseline (Day 1) to Day 30 (Hour 10)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 195 | 191
percentage of participants | 8.7 | 12.6
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.2200, Chi-squared — P-value was adjusted for multiplicity control; Percentage Difference = 3.8, 95% CI 2-sided [-2.3 to 10.0] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline in Mesopic, High-contrast, Binocular DCNVA Letters at Day 30, Hour 0.25
Description: Visual acuity for near (40 cm) target was measured in mesopic conditions using an eye chart. Mesopic condition was defined as low lighting 3.2 to 3.5 cd/m^2 measured at the target. MMRM was used for the analysis.
Time Frame: Baseline (Day 1) to Day 30 (Hour 0.25)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: letters read correctly
Groups:
- Pilocarpine HCl Ophthalmic Solution 1.25%: Participants received one drop of pilocarpine HCl ophthalmic solution 1.25% in each eye, once daily, for up to 30 days.
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution 1.25%
Number analyzed (Participants) | 196 | 193
letters read correctly | 3.9 (0.41) | 6.5 (0.41)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution 1.25%; Test type: Superiority; p < .0001, MMRM — [p-value comment as in outcome 7, analysis 1]; P-value was adjusted for multiplicity control; LS Mean Difference = 2.6, 95% CI 2-sided [1.5 to 3.7], Standard Error of Mean 0.55

10. Secondary Outcome: Percentage of Participants Achieving 20/40 or Better in Photopic, High-contrast, Binocular, DCNVA at Day 30, Hour 3
Description: Visual acuity for near (40 cm) targets was measured in photopic conditions using an eye chart. Photopic condition was defined as high lighting ≥80 cd/m^2 measured at the target.
Time Frame: Day 30 (Hour 3)
Population: ITT Population included all randomized participants. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 198 | 193
percentage of participants | 77.8 | 90.2
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0141, Chi-squared — P-value was adjusted for multiplicity control; Percentage Difference = 12.4, 95% CI 2-sided [5.2 to 19.5] — [estimate comment as in outcome 5, analysis 1]

11. Secondary Outcome: Mean Change From Baseline in Mesopic NVPTQ Satisfaction Score at Day 30, Hour 3
Description: NVPTQ had 12 questions on 4 reading tasks(reading a paragraph from book, excerpts from a newspaper article, portion of a nutrition label, and a section from restaurant menu). Participants completed specific reading tasks under mesopic conditions without any near-vision correction and answered 3 questions for each task, related as 0=I could not read any text due to problems seeing up close,1=poor,2=fair,3=good,4=very good,5=excellent; impact of squinting as 0=No, I did not squint, 1=Yes, squinting helped me read some/all text, 2=Yes, but I still could not read any of the text; and satisfaction as 0=very dissatisfied to 4=very satisfied. NVPTQ Satisfaction Score=(Book testlet+Newspaper testlet+Menu testlet+Nutrition Label testlet)/(testlets with non-missing responses)based on satisfaction items for a total possible score of 0 to 4. Higher scores=better outcomes; a positive change from Baseline indicates higher satisfaction.
Time Frame: Baseline (Day 1) to Day 30 (Hour 3)
Population: ITT Population included all randomized participants. Overall number of participants analyzed is the number of participants with data available for analysis. ANCOVA is used for the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 197 | 192
score on a scale | 0.5 (0.08) | 1.2 (0.08)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p < .0001, ANCOVA — ANCOVA with study intervention group, age group, Baseline binocular DCNVA severity, iris color (brown/non-brown), emmetrope/non-emmetrope, and Baseline domain score as fixed effects; P-value was adjusted for multiplicity control; LS Mean Difference = 0.7, 95% CI 2-sided [0.5 to 1.0], Standard Error of Mean 0.11

12. Secondary Outcome: Mean Change From Baseline in Presbyopia Coping Questionnaire (PICQ) Coping Score at Day 30, Hour 3
Description: PICQ=20 questions about impact experienced by participants due to their problems over past 7 days.PICQ Coping domain had 8 items: 1:Normal-sized text,2:Small-sized text,3:Information on a computer,4:Information on a cell phone,5:Increase font size,6:Use glasses to read close,12:Hold reading materials farther out/closer,13:Squint to read. Each item had response categories:0=never to 4=all the time. Items 3, 4, 5, and 6 had additional response categories with values of 9/10 to indicate the question is not applicable to participant and were assigned missing values.PICQ Coping Score:(Item 1,2 Testlet+Item 3,4 Testlet+Item 5+Item 6+Item 12+Item 13)/non-missing responses to the 6 components of coping score where Items 1,2 Testlet=(Item1+Item2)/non-missing responses to Items 1,2;Items 3,4 Testlet=(Item3+Item4)/non-missing responses to Items 3, 4. Score ranges:0=to least amount of coping to 4=greatest amount of coping. Higher scores=poorer outcome; a negative change from Baseline=improvement.
Time Frame: Baseline (Day 1) to Day 30 (Hour 3)
Population: ITT Population included all randomized participants. Overall number of participants analyzed is the number of participants with data available for analysis. ANCOVA was used for the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 197 | 193
score on a scale | -0.5 (0.06) | -0.9 (0.06)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0002, ANCOVA — [p-value comment as in outcome 11, analysis 1]; P-value was adjusted for multiplicity control; LS Mean Difference = -0.4, 95% CI 2-sided [-0.5 to -0.2], Standard Error of Mean 0.08

13. Secondary Outcome: Mean Change From Baseline in PICQ Impact Score at Day 30, Hour 3
Description: PICQ had 20 questions about impact experienced by participants due to their problems seeing up over past 7 days. Impact domain of PICQ has 6 items:Item9:Rely on others,Item15:rest eyes,Item16:Feel older,Item17:Feel self-conscious,Item19:Take longer to complete task,Item20:Inconvenient.First 5 impacts items include response ranges from 0=never to 4=all of time. Item20 ranged from 0=Not at all,to 4=Extremely. Item9 included an additional response category, labeled with value of 9 to indicate question is not applicable because participant did not have opportunity to experience impact responses are assigned missing values. PICQ Impacts Score=[(Items 9+15+16&17 Testlet+Item19+Item20)/(nonmissing responses to 5 components of impacts score)] where Items 16&17 Testlet=(Items16+17)/non-missing responses to Items16 and 17. PICQ Impact score ranged 0-4, 0=least amount of impacts,4=greatest amount of impacts. Higher scores correspond to poorer outcomes; negative change from Baseline=improvement.
Time Frame: Baseline (Day 1) to Day 30 (Hour 3)
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 197 | 193
score on a scale | -0.4 (0.06) | -0.7 (0.06)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0002, ANCOVA — [p-value comment as in outcome 11, analysis 1]; P-value was adjusted for multiplicity control; LS Mean Difference = -0.3, 95% CI 2-sided [-0.4 to -0.2], Standard Error of Mean 0.07

ADVERSE EVENTS:
Time Frame: First dose of study drug intervention to within 30 days after last dose (Up to 60 days)
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/215 | 0/212
Serious Adverse Events (participants affected / at risk) | 2/215 | 0/212
Other Adverse Events (participants affected / at risk) | 25/215 | 58/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=215) | Pilocarpine HCl Ophthalmic Solution (N=212)
Dysphagia (Gastrointestinal disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=215) | Pilocarpine HCl Ophthalmic Solution (N=212)
Headache (Nervous system disorders) | 11 | 33
Conjunctival hyperaemia (Eye disorders) | 11 | 15
Vision blurred (Eye disorders) | 1 | 13
Eye pain (Eye disorders) | 3 | 12

LIMITATIONS AND CAVEATS:
DCNVA measurements at 1 site were not conducted correctly at the screening and baseline visits; all participants from this site were excluded from efficacy analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT03857542/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT03857542/SAP_001.pdf